CLINICAL TRIAL: NCT03753386
Title: Identification of Respiratory Profiles From Nasal Pressure Signals
Acronym: IPR-SAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Collaborators: SRETT (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-A01999-46
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): Subjects not presenting any pulmonary pathology that will follow the intervention Oxygen therapy simulation.
  Interventions: Other: Oxygen therapy simulation

INTERVENTIONS:
Other: Oxygen therapy simulation — The intervention consists of reproducing oxygen therapy situations in healthy individuals by replacing oxygen bottles with bottles of air. A TeleOx® device will be placed on the circuit between the source and the nasal cannula for respiratory signals recording.
  The intervention will last 30 minutes, containing the following activities in the given order:
  * rest (9 minutes);
  * drinking water (1 minute);
  * rest (1 minute);
  * coughing (1 minute);
  * rest (1 minute);
  * reading aloud (1 minute);
  * rest (1 minute);
  * breathing by the mouth (1 minute);
  * rest (1 minute);
  * exercising (running) (3 minutes) and
  * rest (10 minutes)
  Recordings will be retrieved after each test.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic respiratory disease caused by smoking and associated with significant morbidity due to recurrent exacerbations or even hospitalizations. It is one of the leading causes of death in rich countries.

Early detection of exacerbations of the disease is thus an economic and public health issue in the world. Finding tools for automatic and early detection of an exacerbation is the subject of the study. A continuous analysis of the frequency and shape of the patients' breathing will be used.

As a first step in this study, investigators want to measure the frequency and shape of breathing in healthy subjects as they execute standard activities. These activities include resting, drinking, coughing, speaking, breathing through the mouth, physical exercise and recuperation.

ELIGIBILITY:
Inclusion Criteria:

* Age of majority
* Health volunteers

Exclusion Criteria:

* Pregnancy
* Age of minority
* Protected adult
* Person deprived of liberty
* Respiratory pathology
* Non affiliation to the health care system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Pressure | 10 Hz for 30 minutes
  The monitoring device used records the nasal pressure from users at 10 Hz (one measure every 0.1 seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Gonzalez-Bermejo, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- INSERM-UPC UMR_S 1158, Service de Pneumologie et Réanimation, GH Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Pegoraro JA, Lavault S, Wattiez N, Similowski T, Gonzalez-Bermejo J, Birmele E. Machine-learning based feature selection for a non-invasive breathing change detection. BioData Min. 2021 Jul 18;14(1):33. doi: 10.1186/s13040-021-00265-8. PMID 34275469